CLINICAL TRIAL: NCT03281759
Title: Effects of Transcranial LED Therapy on the Cognitive Rehabilitation for Diffuse Axonal Injury Due to Severe Acute Traumatic Brain Injury: Randomized Clinical Trial.
Brief Title: Transcranial LED Therapy for Severe Acute Traumatic Brain Injury
Acronym: LED-TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15425
Record Dates: First submitted 2017-09-04; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Diffuse Axonal Brain Injury; Traumatic Brain Injury
Keywords: Brain Injuries, Traumatic;; Diffuse Axonal Injury; Low-Level Light Therapy; Neurologic Manifestations; Quality of Life; Rehabilitation
MeSH Terms: conditions — Brain Injuries, Diffuse; Brain Injuries, Traumatic; Diffuse Axonal Injury; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Coil Helmet (Active Comparator): The patients will undergo 18 sessions (627 nm, 70 mW/cm2, 10 J/cm2) at four points of the frontal and parietal region for 30 s each, totaling 120 s three times per week for 6 weeks, lasting 30 minutes of transcranial LED stimulation.
  Interventions: Device: Transcranial LED Therapy (Active coil helmet)
- Inactive Coil Helmet (Placebo Comparator): The patients assigned to this group will undergo 18 sessions of transcranial LED but with an inactive coil, which will not generate LED emissions.
  Interventions: Device: Transcranial LED Therapy (Inactive coil helmet)

INTERVENTIONS:
Device: Transcranial LED Therapy (Active coil helmet) — The patients will undergo 18 sessions of repetitive transcranial LED stimulation.
  Arms: Active Coil Helmet
Device: Transcranial LED Therapy (Inactive coil helmet) — The patients assigned to this group will undergo 18 sessions of transcranial LED but with an inactive coil, which will not generate LED emissions, only a similar red light color.
  Arms: Inactive Coil Helmet

SUMMARY:
The purpose of this study is to evaluate early and delayed effects of Transcranial LED Therapy (TCLT) and determinate whether this therapy is effective for cognitive rehabilitation of Diffuse Axonal Injury patients after Traumatic Brain Injury.

DETAILED DESCRIPTION:
This is a randomized clinical trial of patient with diffuse axonal injury (DAI) secondary to severe Traumatic Brain Injury in its acute stage (less than 8h). It will be recruited thirty adult patients who will receive thirty minutes at three times per week for 6 weeks (18 sessions) of transcranial stimulation. Fifteen of them will be stimulated with LED helmet and the rest with a sham helmet identical to the LED one, but only with a similar red light emission. Patient who meet inclusion criteria will be assessed with Glasgow Outcome Scale Extended (GOS-E) evaluation in at least five different periods (Admission, before and after each stimulation, and at 3 and 6 months later in outpatient followup).

ELIGIBILITY:
Inclusion Criteria:

1) Patient victims of Traumatic Brain Injury with Glasgow Coma Scale ≤8 on admission:

1. Head CT scan showing diffuse axonal lesion.
2. CT scan without focal surgical lesions (Marshall I and II) and no signs of intracranial hypertension.
3. Transcranial Doppler and optic nerve sheath US with no signs of intracranial hypertension.
4. Admission less than 8 hours of trauma.

Exclusion Criteria:

1. History of drug or narcotic abuse.
2. Emergence of surgical lesions or signs of intracranial hypertension in followup CTs.
3. Transcranial Doppler or optic nerve sheath US presenting signs of intracranial hypertension.
4. Psychiatric disorders.
5. Injury severity score ≥3, according to the Abbreviated Injury Scale

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of early and delayed functional outcome measured by Glasgow Outcome Scale Extended (GOSE). | Before stimulation and 1, 3 and 6 months after first stimulation
  Evaluation of improvement of early and delayed functional outcome measured by Glasgow Outcome Scale Extended (GOSE) after stimulation in comparison to the placebo group.

SECONDARY OUTCOMES:
Improvement effects of transcranial LED in followup images measured by Marshall computed tomography scale and Adams grading scale for diffuse axonal injury. | Before stimulation and 1, 3 and 6 months after first stimulation
  Evaluation of early and delayed effects of Transcranial LED Therapy (TCLT) to improve followup computed tomography or magnetic resonance of DAI patients after Traumatic Brain Injury, measured by Marshal computed tomography scale, Adams grading scale for diffuse axonal injury and a protocol published by Hamdeh et al. (doi: 10.1089/neu.2016.4426) which graduates the magnitude of diffuse axonal lesion.
Hemodynamic improvement effect of transcranial LED measured by transcranial doppler (systolic and diastolic velocity of the left middle cerebral and basilar arteries, and the pulsatility index and resistance index values). | Before stimulation and 1, 3 and 6 months after first stimulation
  Improvement evaluation of effects of LED therapy in hemodynamic change through transcranial doppler, measuring systolic and diastolic velocity of the left middle cerebral and basilar arteries, and the pulsatility index and resistance index values.

CONTACTS AND LOCATIONS:
Overall Officials: Wellingson S Paiva, PhD, Study Chair — University of Sao Paulo General Hospital; Joao G Santos, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Santos JGRPD, Zaninotto ALC, Zangaro RA, Carneiro AMC, Neville IS, de Andrade AF, Teixeira MJ, Paiva WS. Effects of transcranial LED therapy on the cognitive rehabilitation for diffuse axonal injury due to severe acute traumatic brain injury: study protocol for a randomized controlled trial. Trials. 2018 Apr 24;19(1):249. doi: 10.1186/s13063-018-2632-5. PMID 29690927